CLINICAL TRIAL: NCT01007669
Title: Effects of Specified Work Site Physical Activity Intervention on Musculoskeletal Disorders Among Employees With Physical Heavy Work
Brief Title: Effects of Specified Work Site Physical Activity Intervention Among Employees With Physical Heavy Work
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bibi Gram (Other)
Responsible Party: Sponsor-Investigator, Bibi Gram, Ph.D student, University of Southern Denmark
Organization: University of Southern Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: s-20090058
Record Dates: First submitted 2009-11-03; First posted 2009-11-04 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2013-02

CONDITIONS: Musculoskeletal Diseases
Keywords: Physical activity
MeSH Terms: conditions — Musculoskeletal Diseases; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Reference (Active Comparator): Health check only
  Interventions: Behavioral: Health check only
- Intervention (Experimental): Physical activity and Health check
  Interventions: Behavioral: Physical activity and Health check

INTERVENTIONS:
Behavioral: Physical activity and Health check — Strength training, aerobic capacity training.
  Arms: Intervention
Behavioral: Health check only — Health check
  Arms: Reference

SUMMARY:
The purpose of this study is to evaluate the effect of specified worksite physical-activity interventions on musculoskeletal disorders in an industry with physical heavy workload.

DETAILED DESCRIPTION:
Studies regarding company adjusted intervention have shown positive effects regarding work related neck and shoulder symptoms among workers with monotonous repetitive work. However, limited research is available on physical exercise intervention among workers with physically heavy work. This study introduces a new intervention concept to treat and prevent musculoskeletal disorders including individually and health check based exercise intervention.

The aim of this randomized controlled intervention project is

1. Through Health check to outline the extent musculoskeletal disability in workers with heavy work load in relation to physical and metabolic fitness. Includes is also assessment of physical general activity and working conditions.
2. To evaluate the effect of individual adjusted exercise programs on muscle strength, aerobic capacity, musculoskeletal disability, pain, work ability and sick absenteeism

ELIGIBILITY:
Inclusion Criteria:

* Constructions workers, working for more than 20 hours pr week, Physical heavy work tasks (in Danish: brolæggere, rørlæggere, mekanikere)

Exclusion Criteria:

* Workers with flexible job i.e. for people with a reduced ability to work

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2009-08; Primary Completion 2010-12 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
muscle strength | 3 months
Aerobic capacity | 3 months

SECONDARY OUTCOMES:
Questionnaire | 1 year
Health Check | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Bibi Gram, M.Sc.,PT, Principal Investigator — University of Southern Denmark
Locations (1):
- University of Southern Denmark, Odense, Denmark

REFERENCES:
- [Derived] Gram B, Westgate K, Karstad K, Holtermann A, Sogaard K, Brage S, Sjogaard G. Occupational and leisure-time physical activity and workload among construction workers - a randomized control study. Int J Occup Environ Health. 2016 Jan;22(1):36-44. doi: 10.1080/10773525.2016.1142724. Epub 2016 Apr 21. PMID 27097799
- [Derived] Holtermann A, Jorgensen MB, Gram B, Christensen JR, Faber A, Overgaard K, Ektor-Andersen J, Mortensen OS, Sjogaard G, Sogaard K. Worksite interventions for preventing physical deterioration among employees in job-groups with high physical work demands: background, design and conceptual model of FINALE. BMC Public Health. 2010 Mar 9;10:120. doi: 10.1186/1471-2458-10-120. PMID 20214807